CLINICAL TRIAL: NCT00843440
Title: Efficacy and Safety of Bevacizumab for the Treatment Hemorrhagic Hereditary Telangiectasia (HHT) Associated With Severe Hepatic Vascular Malformations. Phase II Study.
Acronym: METAFORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008.510/11
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhagic Hereditary Telangiectasia
Keywords: Antiangiogenic therapies; Bevacuzimab; Hemorrhagic Hereditary Telangiectasia (HHT) with severe liver involvement
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Study using a Gehan design, 7 patients will be included in the first phase and 18 additional patients will enter the second phase.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 5 mg / kg every 14 days with a total of 6 injections.A two-phase Gehan method will be used with a first phase designed to eliminate a non effective treatment quickly and a second phase allowing assessment of efficacy.
  Other Names: AVASTIN

SUMMARY:
The efficacy of anti-VEGF treatments such as Bevacizumab in cases of HHT can be considered because of the molecular mechanisms implied in angiogenesis and HHT, as well as the mechanisms of action of this type of treatment. Two articles that have recently reported spectacular improvement thanks to Bevacizumab in patients with HHT complicated with severe liver involvement and cardiac effects support us in this sense.

Up to now, the only treatment recommended in the severe hepatic forms of HHT is a liver transplant, the disadvantages of which are both multiple and well known: long waiting lists, surgical morbidity and mortality, immunosuppressive treatment for life. Furthermore, treatment with Bevacizumab is not a contraindication, should the drug be ineffective, for a subsequent liver transplant if necessary.

ELIGIBILITY:
Inclusion Criteria:

* General criteria:

  * Age ≥ 18 years and < 70 years
  * Subjects must have given their free and enlightened consent and have signed the consent form.
* HHT related criteria

  * Patients monitored for clinically confirmed HHT disease.
  * Patients with severe liver involvement in relationship with the HHT disease
  * Patients with a high cardiac output on ultrasound.
* Associated disease related criteria

  * Blood: neutrophil ≥ 1.0x109 / L and platelets ≥ 100x109 / L.
  * INR (International Normalized Ratio) ≤ 1.5 (except for patients on anticoagulants) and TCA ≤ 1.5 x upper limit of the standard laboratory
  * Renal function: creatinine ≤ 1.25 x upper limit of the standard laboratory. Patients who proteinuria to strip ≥ 2 + will have control of the Proteinuria of 24 hours to be ≤ 1g / 24 hours

Exclusion Criteria:

* • General criteria
* Women who are pregnant or liable to become pregnant in the course of the trial.
* Patients who have reached their majority but who are protected by the terms of the law (French public health code).
* Refusal to give enlightened consent.
* Patients who are not affiliated to a health insurance regime

  • Criteria for the medical history
* Patients in whom the diagnosis of HHT disease has not been confirmed.
* The presence of atrial fibrillation on the electrocardiogram at the inclusion.
* The presence of cerebral arteriovenous malformations on the angioMRI done in the year prior to inclusion.
* Existence of diverticulitis of the colon or sigmoid
* Thrombosis within 6 months before inclusion
* Infectious disease treated by antibiotics and unresolved at inclusion.
* Patients with blood pressure that is not being controlled at the time of inclusion (systolic blood pressure> 150 mmHg and / or diastolic> 100 mmHg) with or without treatment. Patients who have high blood pressure can be included when the blood pressure numbers have been standardized by appropriate medical treatment.

  • Surgical criteria
* Major surgery (including open biopsy) or severe trauma within 28 days preceding the start of treatment.

  • Medical treatments
* Current or recent use of non steroidal anti-inflammatory drugs or antiplatelet therapy 10 days before the first administration of Bevacizumab.
* Use of oral or parenteral anticoagulants or thrombolytic agents within 28 days preceding inclusion (anticoagulants given prophylactically are permitted).
* Participation in another clinical trial within 28 days preceding inclusion.
* Vaccination with live vaccines or against yellow fever during the treatment period.
* Administration of phenytoin (Di-hydan ® DILANTIN ®) during the treatment period.

  • Allergy
* Hypersensitivity to the active substance or any of its excipients.
* Hypersensitivity to products made from Chinese hamster ovary (CHO) cells or to any other human or humanized recombinant antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
cardiac output measured at 3 months | 3 months

SECONDARY OUTCOMES:
Evaluation at 6 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Dupuis-Girod S, Ginon I, Saurin JC, Marion D, Guillot E, Decullier E, Roux A, Carette MF, Gilbert-Dussardier B, Hatron PY, Lacombe P, Lorcerie B, Riviere S, Corre R, Giraud S, Bailly S, Paintaud G, Ternant D, Valette PJ, Plauchu H, Faure F. Bevacizumab in patients with hereditary hemorrhagic telangiectasia and severe hepatic vascular malformations and high cardiac output. JAMA. 2012 Mar 7;307(9):948-55. doi: 10.1001/jama.2012.250. PMID 22396517
- See also: Related Info — http://www.rendu-osler.fr